CLINICAL TRIAL: NCT06183385
Title: Detection of Specific Salivary Proteins by Immunoaffinity and Mass Spectrometry
Brief Title: Detection of Saliva by Immunoaffinity and Mass Spectrometry
Acronym: SIMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL23_0098
Record Dates: First submitted 2023-08-18; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Sexual Assault
Keywords: saliva; proteins; biomarkers; mass spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saliva (Other): Collection of two saliva samples (approx. 1.5 to 2 mL each) by passive drooling in healthy volunteers
  These samples will be centrifuged and the supernatant collected.
  Interventions: Other: Saliva collection; Other: IP-LC-MS/MS : immunoprecipitation enrichment with liquid chromatography coupled to tandem mass spectrometry
- Vaginal secretions (Other): In order to be as close as possible to real life, two vaginal swabs (introduced through the vaginal orifice over a length of 2 to 3 cm) will be taken with a sterile dry swab during the gynecological examination (prior to endovaginal ultrasound or any other endovaginal procedure) of patients included in the Reproductive Medicine Service.
  Interventions: Other: Vaginal secretion collection; Other: IP-LC-MS/MS : immunoprecipitation enrichment with liquid chromatography coupled to tandem mass spectrometry

INTERVENTIONS:
Other: Saliva collection — Collection of 2 samples of 1.5 to 2mL of saliva by passive salivation in healthy volunteers
  Arms: Saliva
Other: Vaginal secretion collection — Collection of vaginal secretions with 2 dry swabs in women
  Arms: Vaginal secretions
Other: IP-LC-MS/MS : immunoprecipitation enrichment with liquid chromatography coupled to tandem mass spectrometry — sample preparation and analysis :
  * Impregnation of the tips (absorbent cotton) of sterile dry swabs and vaginal swabs with controlled quantities of saliva.
  * Immunocapture of salivary proteins of interest (histatin type 1, cystatin D, PRPs) by protein A affinity purification
  * LC-MS/MS analysis of eluted purified peptides (Multiple Reaction Monitoring mode)
  Dilutions will be made from 10 to 10 (1/10, 1/100, 1/1000...), then after reaching a detectability threshold, specified by a second more precise analysis (e.g. if no signal at 1/1000, analysis at 1/500 then 1/250 etc.). Analytical sensitivity will be tested on three samples of each type (salivary, vaginal, vaginal + semen) to ensure reproducibility of results.
  Operators, unaware of the presence of saliva in the samples, will then carry out saliva-specific protein detection analysis using the IP-LC-MS/MS method.

SUMMARY:
The identification of saliva in genital area during a criminal investigation can be a critical component in the prosecution of a sexual assault in France, as non-consensual oral-genital intercourses have been considered as crimes since 2021.The development of highly specific methods for saliva detection is therefore crucial as the commonly employed screening methods lack specificity. Protein mass spectrometry has proven to be a sensitive and specific method but is particularly time consuming. A faster and more sensitive hybrid approach using automated immunoaffinity mass spectrometry (IP-LC-MS/MS) has been recently developed and has been found to be particularly performant for the detection of a seminal fluid protein (semenogelin), allowing a high-throughput seminal fluid identification in semen samples. Like semenogelin, specific salivary proteins such as histatin type 1, cystatin D or proline-rich proteins (PRPs) could be detected using this promising approach, which has never been tested on saliva samples. In collaboration with the Clinical Proteomics Platform and the Department of Reproductive Medicine of the University Hospital of Montpellier, we aim to develop a protocol for the detection of specific saliva proteins by IP-LC-MS/MS in sexual assault-type samples.

DETAILED DESCRIPTION:
Each participant will be contacted by a phone call the day before the visit, to present for a presentation of the study.The day of the visit, two types of samples will be collected :

* Saliva samples: on healthy volunteers in the Department of Legal Medicine (2 samples of 1.5 - 2 mL are collected for each volunteer).
* Vaginal samples : on women consulting in the Department of Reproductive Medicine (2 dry swabs on each patient). 2 groups, One group with vaginal secretion fluid samples only, and one group with vaginal secretion fluid + sperm samples.

ELIGIBILITY:
Inclusion Criteria:

Saliva Samples

* Men and women aged 18 or more

Vaginal samples :

* Women aged 18 or more
* No unprotected vaginal sexual intercourse during the 10 days prior to the visit (group 1)
* Unprotected vaginal sexual intercourse with ejaculation in the 24 hours prior to the visit (group 2)

Exclusion Criteria:

Saliva Samples :

* Active pathology of the saliva glands (infection, tumor)
* Unprotected oral-genital sexual intercourse in the 24 hours prior to the visit
* Failure to obtain written informed consent after a reflection period
* Pregnant or breast feeding women
* Adult protected by law or under guardianship or curatorship
* No affiliation to the French Social Security System or no benefit from such a system

Vaginal Samples :

* Oral-genital sexual intercourse (cunnilingus) in the 24 hours prior to the visit
* Failure to obtain written informed consent after a reflection period
* Pregnant or Breastfeeding women
* Adult protected by law or under guardianship or curatorship
* No affiliation to the French Social Security System or no benefit from such a system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reproducibility between saliva samples | 3 months
  Intra-assessor agreement on saliva samples, which involves testing the first sample and retesting the second sample
  The study's primary endpoint will be to measure the reliability of the protocol, consisting of reproducibility or intra-assessor agreement,for the detection of specific salivary proteins (histatin type 1, PRPs, cystatin D) using the IP-LC-MS/MS method on adult saliva samples.
  Intra-assessor agreement (test/retest) will be measured by their means +/- standard deviation.
  Several analyses (between 3 or 4) on the same sample will be carried out to determine whether the results are identical
Intermediate fidelity between technicians on saliva samples | 3 months
  Inter-assessor agreement(Cohen's kappa coefficient) on saliva samples, which involves testing several samples by at least 2 different technicians
  The study's primary endpoint will be to measure the reliability of the protocol, consisting of intermediate fidelity or inter-assessor agreement (Cohen's kappa coefficient) for the detection of specific salivary proteins (histatin type 1, PRPs, cystatin D) using the IP-LC-MS/MS method on adult saliva samples.
  The kappa coefficient gives a score ranging from 0 to 1. If the coders totally agree, κ = 1. If they totally disagree (or agree due solely to chance), κ ≤ 0.

SECONDARY OUTCOMES:
Reproducibility between vaginal samples soaked with saliva | 3 months
  Intra-assessor agreement on vaginal samples soaked with saliva
  The secondary endpoints, will consist of repeating the primary endpoints (i.e. reproducibility and intermediate fidelity) on the vaginal samples impregnated with sperm or not.
  Again, the same sample will be tested several times (between 3 or 4) to see if the results come back similar.
Intermediate fidelity between technicians on vaginal samples soaked with saliva | 3 months
  : Inter-assessor agreement (Cohen's kappa coefficient) on vaginal samples soaked with saliva
  The secondary endpoints, will consist of repeating the primary endpoints (i.e. reproducibility and intermediate fidelity) on the vaginal samples impregnated with sperm or not.
  The kappa coefficient gives a score ranging from 0 to 1. If the coders totally agree, κ = 1. If they totally disagree (or agree due solely to chance), κ ≤ 0.
Analytical Sensibility | 3 months
  Lowest saliva concentration (µL) detected by the method on saliva samples and on vaginal samples soaked with saliva in controlled condition
Diagnostic sensibility | 3 months
  Analysis of saliva samples and vaginal samples soaked with saliva in controlled condition, to determine the rate of detection of true positives and false negatives
Diagnostic specificity | 3 months
  Analysis of vaginal samples and dry samples in controlled condition, to determine the rate of false positives and true negatives.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Antoine PEYRON, PI, Study Director — University Hospital, Montpellier
Locations (1):
- PEYRON, Montpellier, France

REFERENCES:
- [Background] LOI n°2021-478 du 21 avril 2021 visant à protéger les mineurs des crimes et délits sexuels et de l'inceste. JORF n°0095 du 22 avril 2021. Texte n°4
- [Background] Wornes DJ, Speers SJ, Murakami JA. The evaluation and validation of Phadebas(R) paper as a presumptive screening tool for saliva on forensic exhibits. Forensic Sci Int. 2018 Jul;288:81-88. doi: 10.1016/j.forsciint.2018.03.049. Epub 2018 Apr 20. PMID 29734053
- [Background] Vandenberg N, van Oorschot RA. The use of Polilight in the detection of seminal fluid, saliva, and bloodstains and comparison with conventional chemical-based screening tests. J Forensic Sci. 2006 Mar;51(2):361-70. doi: 10.1111/j.1556-4029.2006.00065.x. PMID 16566772
- [Background] Blanchard Muller M., Baccino E., Peyron P.A. Détection de traces salivaires dans le cadre d'agressions sexuelles : intérêt de l'utilisation d'une méthode immuno-chromatographique rapide (RSID-SalivaTest®) selon un protocole simplifié. Rev Médecine Légale 2023.
- [Background] Davidovics R, Saw YL, Brown CO, Prinz M, McKiernan HE, Danielson PB, Legg KM. High-throughput seminal fluid identification by automated immunoaffinity mass spectrometry. J Forensic Sci. 2022 May;67(3):1184-1190. doi: 10.1111/1556-4029.14975. Epub 2022 Jan 13. PMID 35023573
- [Background] Sato H, Nakajima D, Ishikawa M, Konno R, Nakamura R, Ohara O, Kawashima Y. Evaluation of the Suitability of Dried Saliva Spots for In-Depth Proteome Analyses for Clinical Applications. J Proteome Res. 2022 May 6;21(5):1340-1348. doi: 10.1021/acs.jproteome.2c00099. Epub 2022 Apr 21. PMID 35446574
- [Background] Yang H, Zhou B, Deng H, Prinz M, Siegel D. Body fluid identification by mass spectrometry. Int J Legal Med. 2013 Nov;127(6):1065-77. doi: 10.1007/s00414-013-0848-1. Epub 2013 Mar 24. PMID 23525663
- [Background] Brown CO, Robbins BL, McKiernan HE, Danielson PB, Legg KM. Direct seminal fluid identification by protease-free high-resolution mass spectrometry. J Forensic Sci. 2021 May;66(3):1017-1023. doi: 10.1111/1556-4029.14646. Epub 2020 Dec 8. PMID 33289932
- [Background] Legg KM, Powell R, Reisdorph N, Reisdorph R, Danielson PB. Discovery of highly specific protein markers for the identification of biological stains. Electrophoresis. 2014 Nov;35(21-22):3069-78. doi: 10.1002/elps.201400125. Epub 2014 Oct 1. PMID 25070728
- [Background] Van Steendam K, De Ceuleneer M, Dhaenens M, Van Hoofstat D, Deforce D. Mass spectrometry-based proteomics as a tool to identify biological matrices in forensic science. Int J Legal Med. 2013 Mar;127(2):287-98. doi: 10.1007/s00414-012-0747-x. Epub 2012 Jul 29. PMID 22843116
- [Background] Illiano A, Arpino V, Pinto G, Berti A, Verdoliva V, Peluso G, Pucci P, Amoresano A. Multiple Reaction Monitoring Tandem Mass Spectrometry Approach for the Identification of Biological Fluids at Crime Scene Investigations. Anal Chem. 2018 May 1;90(9):5627-5636. doi: 10.1021/acs.analchem.7b04742. Epub 2018 Apr 13. PMID 29579379
- [Background] Legg KM, Powell R, Reisdorph N, Reisdorph R, Danielson PB. Verification of protein biomarker specificity for the identification of biological stains by quadrupole time-of-flight mass spectrometry. Electrophoresis. 2017 Mar;38(6):833-845. doi: 10.1002/elps.201600352. Epub 2017 Jan 30. PMID 27943336
- [Background] de Beijer RP, de Graaf C, van Weert A, van Leeuwen TG, Aalders MCG, van Dam A. Identification and detection of protein markers to differentiate between forensically relevant body fluids. Forensic Sci Int. 2018 Sep;290:196-206. doi: 10.1016/j.forsciint.2018.07.013. Epub 2018 Jul 24. PMID 30071450
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/29734053/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/16566772/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35023573/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/35446574/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/23525663/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/34311288/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/25070728/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/22843116/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/29579379/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/27943336/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/30071450/